CLINICAL TRIAL: NCT05864482
Title: The Effect of Psychosocial Nursing Interventions on Sleep, Anxiety and Delirium in Patients Undergoing Open Heart Surgery
Brief Title: Psychosocial Nursing Interventions on Sleep, Anxiety and Delirium in Patients Undergoing Open Heart Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, FİRDEVS EBRU ÖZDEMİR, Specialist Nurse, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Interventional
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Delirium
Keywords: psychosocial nursing interventions; sleep; anxiety; delirium
MeSH Terms: conditions — Delirium; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Brief Cognitive behavioral therapy intervention will be interviewed by the researcher as part of psychosocial care, with two sessions pre-operative and two post-operative sessions. In the postoperative period, an eye mask and ear plug will be applied to the patient by the researcher on the 3rd and 4th days of the short CBT post-op and between 23:00 and 07:00 at night. Visual Analogue Scale, State Anxiety Inventory, Richmond Agitation-Sedation Scale, Confusion Evaluation Scale in Intensive Care, Richard Campbell Sleep Quality Scale, Daily Follow-up Form will be applied after open heart surgery.
  Interventions: Other: Psychosocial nursing intervention
- Control (No Intervention): Patients who meet the research criteria and agree to participate in the study will be informed about the research process (purpose of the research, assignment to the intervention and control group, etc.), written informed consent and contact information of the patients will be obtained, and the contact information of the researcher will be given to the patient. Only routine nursing care will be given to the patient. will be applied by the researcher

INTERVENTIONS:
Other: Psychosocial nursing intervention — The sessions were planned to be at least 45 minutes in a time suitable for the groups, with the bed curtains drawn if possible. Session 1: The purpose of this session; Brief CIS information will be provided. Session 2: The session starts with mood control of individuals. It is discussed whether they have experienced an event that occupies their minds and is likely to affect their illness. Session 3: It starts with mood control of individuals. They are asked if there is anything from the places where the guests are. Cognitive reviews are reviewed. It aims to describe recent stressful observations, negative automatic outcome descriptions, and evaluation of such experiences. 4.Session: The session starts with the mood control of the patient. It is discussed whether the patient has experienced an event that occupies his mind. Continuous analysis of negative thoughts and review of cognitive techniques and coping mechanisms are provided.
  Arms: Experimental

SUMMARY:
The goal of this study is to determine the effects of psychosocial nursing interventions applied to a patient with cardiac surgery on sleep quality, anxiety and delirium.

Are psychosocial nursing interventions applied to a patient with cardiac surgery effective in preventing delirium?

Are psychosocial nursing interventions applied to a patient with cardiac surgery effective on sleep quality?

Are psychosocial nursing interventions applied to a patient with cardiac surgery effective on the level of anxiety?

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) are among the most common leading causes of death worldwide. Among cardiovascular diseases, coronary artery disease (CAD) is an important health problem that is the most common and causes death. Medical treatment and revascularization have an important place among the treatment methods of CAD. Revascularization is performed with stenting and/or coronary artery bypass surgery (CABC) according to the patient's clinic and coronary artery lesions. CABC in the world is generally performed using open heart surgery heart-lung pump. Open heart surgeries aim to reduce mortality and morbidity and improve quality of life. Despite all the scientific and technological developments in open heart surgery, some patients may have physical and psychological recovery problems. The patients' own heart problems and information about the heart from the environment; It causes intense fear of death and anxiety in some of the individuals who will undergo heart surgery in the pre- and post-operative period. Revealed in this process; Persistent symptoms may occur due to anxiety, stress, depression, pain, fatigue, and sleep disorders. It may not always be possible to effectively eliminate these complications with pharmacological treatments. Cognitive-Behavioral Therapy (CBT) can be an alternative to pharmacological treatment, and it can be applied together with drugs to help resolve problems. CBT is a proven and accepted psychotherapeutic method based on clinical experience, theory and research. There are three categories of CBT. The first is the origin of behavioral therapy; The second is based on theories about thoughts and their effects on the body, emotions, and actions (cognitive therapy), while the third category of CBT (acceptance and commitment therapy), metacognitive therapy, and mindfulness-based therapy are based on acceptance. The focus in cognitive therapy is on which thought and behavioral patterns of the patient can create and perpetuate existing problems and affect functional levels. It can manage the level of depression and anxiety by changing thought and behavior patterns. One of the common neurofunctional complications after cardiovascular surgery is delirium. Delirium manifests as a disturbance of consciousness and attention accompanied by changes in cognitive function or perceptual impairment. Delirium is characterized by acute onset and recurrent fluctuations. Patients who need constant monitoring and care in the intensive care unit after open heart surgery find themselves surrounded by medical and technological equipment. Many factors such as sedation, environmental factors, illness and mechanical ventilation affect the incidence of anxiety and delirium by causing sleep disturbance and confusion in the concepts of day and night in patients hospitalized in the intensive care unit. It is assumed that reducing environmental factors such as excessive noise and alarms and exposure to artificial light in intensive care can improve the patient's sleep quality. In this respect, it is thought that the use of earplugs and eye masks will be effective measures in patients. Considering that the cause of delirium is multifactorial, it is recommended that nurses integrate it into care by reducing pain, providing orientation, meeting sensory motor requirements such as glasses and hearing aids, maintaining biological sleep patterns, and reducing anxiety. In this context, it is thought that CBT and eye mask, ear plug applications, which are non-pharmacological psychosocial nursing interventions, can be used as an independent nursing intervention to improve sleep quality and prevent anxiety and delirium. In addition, melatonin and cortisol hormones both play a role in regulating the sleep-wake cycle. The core area of delirium is represented by the disruption of sleep. In this respect, the post-operative blood melatonin and cortisol levels of the patients will be examined as secondary outcomes of the study.

ELIGIBILITY:
Inclusion Criteria:

Between 15 April - 31 August 2023, Mersin University Hospital cardiovascular surgery service, cardiovascular surgery intensive care unit was admitted,

* over the age of 18,
* Patients who will undergo open heart surgery for the first time,
* Not diagnosed with any psychiatric disease,
* Conscious, cooperative, hemodynamically stable (blood pressure not below 70/50mHg), not on mechanical ventilator
* Patients with a state anxiety scale score of 40 and above,
* Low and medium risk patients evaluated with the European System for Cardiac Operative Risk Evaluation (EuroSkor), the risk scoring system used to predict mortality in the preoperative period in cardiac surgery,
* Literate, with sufficient communication skills and Turkish-speaking
* Those who signed the Informed Consent Form to participate in the study will be included.

Exclusion Criteria:

Between 15 April - 31 August 2023, Mersin University Hospital cardiovascular surgery service, cardiovascular surgery intensive care unit was admitted,

* Emergency patients for whom open heart surgery has not been planned before,
* Diagnosed with dementia,
* Standardized mini mental test (SMMT) below 3 points,
* Has a history of previous cerebrovascular accident (CVO),
* Severe comorbidity
* Patients with a high EuroScore and prolonged mechanical ventilator duration
* Those who do not sign the Informed Consent Form to participate in the study will not be included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in sleep quality on the Richard Campell Sleep Quality Scale at two days | Baseline and two days
  This scale, developed by Richards, is a 6-item scale that measures the depth of night sleep, the time to fall asleep, the frequency of awakening, the time to stay awake when awakened, the quality of sleep, and the noise level in the environment. Each item is evaluated on a chart with numbers from 0 to 100. According to the scale scoring, "0-25" points indicate very bad sleep, while "76-100" points indicate very good sleep. The 6th item, which evaluates the noise level in the environment, is excluded from the scale total score evaluation, and the total score is evaluated over 5 items. As the score of the scale increases, the sleep quality of the patients also increases.
Change from baseline in pain on the Visual Analog Scale at two days | Baseline and two days
  Developed by Price et al. (1983), this scale is one of the commonly used pain measurement tools in health research due to its ease of use and simple structure. The scale consists of a 10 cm ruler on which there is no pain on one end and excruciating pain on the other end, on which the patient marks the pain. The distance between the point where the patient marked the pain and the pain-free interval is measured in cm and recorded. Cline et al., in their study to standardize the VAS, determined that the vertical use of the VAS was better understood by the patients.
Change from baseline in anxiety on the State Anxiety Scale at two days | Baseline and two days
  The State-Trait Anxiety Inventory was developed by Spielberger et al. in 1970 to measure state anxiety and trait anxiety. The Turkish validity and reliability study of the scale was performed by Le Compte and Öner in 1983. The "state anxiety" to be used in this study is the subjective fear that the individual feels due to the stressful situation he is in. The state anxiety scale is an easy-to-apply inventory consisting of 20 questions that the individual can answer himself. The individual is asked to mark one of the statements (1) "not at all", (2) "somewhat", (3) "a lot", and (4) "completely", evaluating how he or she feels "at the moment". If the lowest score that can be obtained at the end of the scale is 20, the highest score is 80. In the evaluation, 0-19 points are interpreted as "no anxiety", 20-39 points as "mild anxiety", 40-59 points as "moderate anxiety", 60-79 points as "severe anxiety" and 80 points as "panic value".

SECONDARY OUTCOMES:
Change from baseline in delirium on the Confusion Evaluation in Intensive Care Scale at two days | Baseline and two days
  It is included in the nursing observations, and that delirium could be diagnosed early in the intensive care unit and treated by taking precautions against complications [37]. The scale consists of four items. Sudden change or fluctuation of consciousness in the first item; In the second item, squeezing the hand in less than 12 letters in the attention assessment test tests the two most important signs of delirium, fluctuations in the level of consciousness and deterioration of attention. In the third item, whether the organization of thought is disrupted is evaluated by following four questions and a simple command. The fourth item is about the assessment of the level of consciousness. According to this scale, in order to diagnose delirium, the first two items and one of the third or fourth items must be positive.
Change from baseline in agitation on the Richmand Sedation Agitation Scale at two days | Baseline and two days
  Sessler and others. It was developed by in 2002 to evaluate sedation status in adult ICU patients. In order to be able to evaluate delirium, first of all, the state of consciousness (wakefulness) should be evaluated. It takes ten different values between (+4) and (-5) on the RASS scale. While the ideal level at which the patient is awake and calm is scored with "0" on the scale, scores up to "+4" indicate the increasing agitation of the patient and scores up to "-5" indicate the patient's increasing level of sedation.

CONTACTS AND LOCATIONS:
Overall Officials: Mualla YILMAZ, PhD, Study Director — Prof. Dr.
Locations (1):
- Firdevs Ebru ÖZDEMİR, Mersin, Yenişehir, Turkey (Türkiye)